CLINICAL TRIAL: NCT03761888
Title: How Nicardipine and Labetalol Affect Cerebral Hemodynamics in Severe Preeclamptic Patients: A Pilot Observational Study
Brief Title: Nicardipine and Labetalol Effects on Cerebral Hemodynamics in Preeclampsia
Acronym: PREMODYM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hopital Antoine Beclere (Other)
Responsible Party: Principal Investigator, Dr Mickaël Soued, Principal Investigator, Hopital Antoine Beclere
Other Study IDs: 2018-A00689-46
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Preeclampsia Severe
MeSH Terms: interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Labetalol: Patients who will receive labetalol in IV route in first intention
  Interventions: Diagnostic Test: optic nerve sheath measurement and transcranial doppler
- Nicardipine: Patients who will receive nicardipine in IV route in first intention
  Interventions: Diagnostic Test: optic nerve sheath measurement and transcranial doppler

INTERVENTIONS:
Diagnostic Test: optic nerve sheath measurement and transcranial doppler — evaluation of cerebral hemodynamics through measurement of systolic and diastolic velocities and PI in middle cerebral artery. Intracranial pressure will be appreciate by optic nerve sheath value

SUMMARY:
Realization of transcranial doppler and optic nerve sheath in severe preeclamptic patients to evaluate the impact of nicardipine and labetalol on cerebral hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Aged up to 18 years
* patient with severe preeclampsia defined by Systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg after 20 weeks of amenorrhea, associated with neurologic troubles, eclampsia of epigastric pain.
* Decision by clinician to introduce an antihypertensive therapy by oral route : either labetalol or nicardipine

Exclusion Criteria:

* history of intracranial expansive processus, surgery or vascular disease
* infectious state on probe placement
* unilateral anophthalmia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with severe preeclampsia and antihypertensive drug administrated by i.v. route
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-11-29 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Change of values obtained by ultrasonography optic nerve sheath measurement from baseline to 2 hours post starting infusion of nicardipine or labetalol. | just before treatment and 2 hours after
  Variation of values will be studied during a 2 hour time period, starting just before administration of either labetalol or nicardipine by i.v. route

SECONDARY OUTCOMES:
variation of diastolic and systolic velocities in middle cerebral artery before and after administration of either labetalol or nicardipine by i.v. route | just before treatment and at 30 minutes to 60 minutes, 2 hours to 3 hours and 6 hours to 8 hours
  values are obtained by transcranial doppler
variation of PI in middle cerebral artery before and after administration of either labetalol or nicardipine by i.v. route | just before treatment and at 30 minutes to 60 minutes, 2 hours to 3 hours and 6 hours to 8 hours
  values are obtained by transcranial doppler
proportion of pathologic PI in middle cerebral artery in each group | just before treatment and at 30 minutes to 60 minutes, 2 hours to 3 hours and 6 hours to 8 hours
  values are obtained by transcranial doppler
proportion of optic nerve sheath up to 5.8 mm in each group | just before treatment and at 30 minutes to 60 minutes, 2 hours to 3 hours and 6 hours to 8 hours
  values are obtained by ultrasonography
values of optic nerve sheath diameter in each group | At 30 minutes to 60 minutes and 6 hours to 8 hours
  values are obtained by ultrasonography

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Béclère, Clamart, France

IPD SHARING:
Plan to Share IPD: No